CLINICAL TRIAL: NCT02755870
Title: A Phase 1 Single-Ascending Dose (SAD) and Multiple- Ascending Dose (MAD) Study of CNM-Au8 in Healthy Male and Female Volunteers
Brief Title: A Phase I SAD and MAD Clinical Trial of CNM-Au8 in Healthy Male and Female Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Clene Nanomedicine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AU8.1000-14-01
Record Dates: First submitted 2016-04-23; First posted 2016-04-29 (Estimated); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Healthy Volunteers - Male and Female
MeSH Terms: interventions — Nanoparticles

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNM-Au8 (Experimental): CNM-Au8 is an orally administered, clean-surface gold nanocrystal suspension drug. It is atomically clean-surface elemental nanocrystals, free of any residual surface chemicals or surface-capping agents.
  CNM-Au8 15, 30, 60, 90mg as an oral suspension
  Interventions: Other: CNM-Au8
- Placebo (Placebo Comparator): Placebo oral suspension which matches the volume of the experimental nanocrystal suspension
  Interventions: Other: Placebo

INTERVENTIONS:
Other: CNM-Au8 — Clene's technology integrates nanotechnology, materials science, plasma conditioning (corona discharge), and hydro-electrocrystallization to create a new nanocatalytic drug class
  Other Names: Nanoparticles, clean surface nanocrystals
  Arms: CNM-Au8
Other: Placebo — Placebo oral suspension which matches the volume of the experimental nanocrystal suspension
  Arms: Placebo

SUMMARY:
This is a Phase 1, First-Time-In-Humans, randomized, placebo-controlled, double-blind, escalating single- and multiple-dose study to evaluate the safety, tolerability, and pharmacokinetics of CNM-Au8 in healthy male and female volunteers. There will be 2 phases to this study: a single ascending dose (SAD) phase and a multiple ascending dose (MAD) phase. The SAD Phase will be conducted first followed by the MAD phase of the study.

DETAILED DESCRIPTION:
SAD Phase:

A total of 8 subjects will be randomly assigned in a 3:1 ratio to receive a single dose of either CNM-Au8 (n=6) or placebo (n=2) at an initial dose level of 15 mg CNM-Au8. Additional cohorts of 8 subjects will be enrolled to investigate escalating single doses of CNM-Au8 at 30, 60, and 90 mg. Cohorts will be balanced by sex with no more than 2/3rd of subjects being of one sex.

MAD Phase:

A total of 12 subjects will be randomly assigned in a 3:1 ratio to receive a multiple dose of either CNM-Au8 (n=9) or placebo (n=3) once daily for 21 days at an initial dose level of 15 mg CNM-Au8. Additional cohorts of 12 subjects will be enrolled to investigate escalating multiple doses of CNM-Au8 at 30, 60, and 90 mg CNM Au8 administered once daily for 21 days. Cohorts will be balanced by sex with no more than 2/3rd of subjects being of one sex.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB) approved informed consent is signed and dated prior to any study-related activities.
* Females will be non-pregnant, non-lactating, or post-menopausal
* All laboratory values at screening fall within normal range or are evaluated as not clinically significant
* Has not consumed and agrees to abstain from taking any dietary supplements or non-prescription drugs
* Has not consumed and agrees to abstain from taking any prescription drugs
* Has not consumed alcohol-containing beverages
* Has not consumed grapefruit or grapefruit juice
* Has not used tobacco- and nicotine-containing products
* Has the ability to understand the requirements of the study and is willing to comply with all study procedures.

Exclusion Criteria:

* Has a history of illicit drug abuse
* Has clinically significant medical or psychiatric history
* Has donated plasma or excessive blood loss
* Prior participation in another clinical trial

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Treatment emergent adverse and serious adverse events | 49 days
  Occurrence of adverse events
Tmax | Single dose and up to 21 days of consecutive daily dosing
  Time to Cmax
CL/F | Single dose and up to 21 days of consecutive daily dosing
  The apparent systemic clearance
t 1/2 | Single dose and up to 21 days of consecutive daily dosing
  Terminal phase half-life
Cmax | Singe dose and up to 21 days of consecutive daily dosing
  Maximum observed plasma concentration

SECONDARY OUTCOMES:
Changes in cytokine levels | Following a single oral dose or multiple oral doses (once daily for 21 consecutive days)
  Immune modulating effects of orally administered CNM-Au8

CONTACTS AND LOCATIONS:
Overall Officials: G.J. Groeneveld, MD, PhD, Principal Investigator — Centre for Human Drug Research
Locations (1):
- Centre for Human Drug Research (CHDR), Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided